CLINICAL TRIAL: NCT04874142
Title: Phase 1 to Evaluate the Safety and Pharmacokinetic Durg-drug Interaction of YYC506-T and YYC506-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYPCT_YYC506_P1_DDI
Record Dates: First submitted 2021-04-20; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: two-cohort, single-sequence, parallel, open label, multiple oral dosing study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Experimental): Two cohort, single sequence
  Interventions: Drug: YYC506-T; Drug: YYC506-T + YYC506-A
- B Group (Experimental): Two cohort, single sequence
  Interventions: Drug: YYC506-A; Drug: YYC506-A + YYC506-T

INTERVENTIONS:
Drug: YYC506-T — single administration
  Arms: A Group
Drug: YYC506-A — single administration
  Arms: B Group
Drug: YYC506-T + YYC506-A — concomotant administration
  Arms: A Group
Drug: YYC506-A + YYC506-T — concomotant administration
  Arms: B Group

SUMMARY:
To evaluate the safety and pharmacokinetics drug-drug interaction of YYC506-T and YYC506-A

DETAILED DESCRIPTION:
Phase 1 to evaluate the safety and pharmacokinetics drug-drug interaction of YYC506-T and YYC506-A. Which is designed as two cohort, single-sequence, paralle, open label, multiple oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 ages healty men
* Over 50.0kg, 18.0kg/m2 ≤ BMI ≤30.0kg/m2
* Men who dont have congenital disease and other cronic disease need to be cared etc.

Exclusion Criteria:

* Men who have congenital liver disease (AST, ALT, CK ≥ 2X ULN)
* Men who have drunken or eatten something including carffeine within 24 hours before etc.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokietic parameters administration: Cmax | Until 48 hours
  YYC506-T, YYC506-A, and concomitant administration Cmax
Pharmacokietic parameters administration: AUC | Until 48 hours
  YYC506-T, YYC506-A, and concomitant administration AUC

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, PhD, Study Chair — ChungBuk National Unviersity Hospital.
Locations (1):
- ChungBuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No